CLINICAL TRIAL: NCT05810805
Title: Measurement and Analysis of Gas Composition in Digestive Tract: a Prospective, Single-center Observational Study
Brief Title: Measurement and Analysis of Gas Composition in Digestive Tract
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xiuli Zuo (Other)
Responsible Party: Sponsor-Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Organization: Shandong University (Other)
Other Study IDs: 2023SDU-QILU-G001
Record Dates: First submitted 2023-02-13; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Inflammatory Bowel Diseases; Irritable Bowel Syndrome; Functional Dyspepsia; Colorectal Neoplasms; Helicobacter Pylori Infection
MeSH Terms: conditions — Inflammatory Bowel Diseases; Irritable Bowel Syndrome; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Control group
  Interventions: Other: gas component of digestive tract
- Imflammtory bowel disease group
  Interventions: Other: gas component of digestive tract
- Irritable bowel syndrome group
  Interventions: Other: gas component of digestive tract
- Colorectal neoplasms group
  Interventions: Other: gas component of digestive tract
- Helicobacter pylori infection group
  Interventions: Other: gas component of digestive tract
- functional dyspepia group
  Interventions: Other: gas component of digestive tract

INTERVENTIONS:
Other: gas component of digestive tract — Analyze the differences in gas components in different segments of the digestive tract in patients with different diseases, and analyze the correlation between specific gases and digestive tract diseases and non-specific symptoms.

SUMMARY:
The purpose of this study is to detect the concentration of various gases，including hydrogen, methane, hydrogen sulfide, nitric oxide in different parts of the digestive tract by a safe and direct method, and to establish a human digestive tract gas profiles. Analyze the differences in gas components in different segments of the digestive tract in patients with different diseases, and analyze the correlation between specific gases and digestive tract diseases and non-specific symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 70 years.
* Patients undergoing endoscopic examination

Exclusion Criteria:

* Patients with serious underlying diseases, such as liver insufficiency, renal insufficiency, immunosuppression, coronary heart disease (angina pectoris or coronary artery stenosis ≥ 75%).
* Patients have history of gastrointestinal surgery
* Patients who failed to complete the endoscopic examination due to various reasons
* Patients Boston score of Bowel preparation≤ 6 points
* Patients who have medication history of probiotics, antibiotics, PPIs and prokinetic drugs in the last 4 weeks
* Patients who combined with thyroid disease and other diseases that affect gastrointestinal motility
* Patients who combined with other risk factors such as mental illness, alcoholism, and drug abuse
* Patients who unable or unwilling to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing endoscopy at Qilu Hospital of Shandong University
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-03-02 (Estimated)

PRIMARY OUTCOMES:
Concentrations of different gas in digestive tract | immediately after the procedure
  Concentrations of H2, CH4, NO and H2S in various parts of digestive tract

SECONDARY OUTCOMES:
Correlation between digestive tract and breath test | Immediately after the procedure
  Correlation between concentration levels of H2, CH4, NO and H2S in various parts of digestive tract and breath test
Differences in concentrations of H2, CH4, NO, and H2S in the digestive tract between patients with different gastrointestinal diseases and normal individuals. | Immediately after the procedure
  The diagnosis of imflammtory bowel disease, irritable bowel syndrome, colorectal neoplasms, helicobacter pylori infection and functional dyspepia refer to Chinese guidelines or expert consensus. The gas sample will be taken through the biopsy port during endoscopy. The concentration of H2, CH4, NO and H2S will be assessed by chemical gas sensor. The measured concentration of H2 and CH4 is one part per million(ppm). For NO and H2S, the measured concentration is one part per billion (ppb). For different disease groups, the difference between the control groups and the disease group will be analyzed with Student's t test or Mann-Whitney U test.
The correlation between the severity of gastrointestinal symptoms and gas concentrations in various parts of the digestive tract. | Immediately after the procedure
  The symptoms will be assessed by Gastrointestinal Symptom-Rating Scale (GSRS) scores. The gas sample will be taken through the biopsy port during endoscopy. The concentration of H2, CH4, NO and H2S will be assessed by chemical gas sensor. The measured concentration of H2 and CH4 is one part per million(ppm). For NO and H2S, the measured concentration is one part per billion (ppb). The Spearman correlation will be used to determine the correlation between the severity of gastrointestinal symptoms and different gas concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China